CLINICAL TRIAL: NCT07150338
Title: Outcome of Use of a Novel Modulator of Oxidative Phosphorylation on Kidney Function in Patients With Chronic Kidney Disease
Brief Title: Outcome of Use of a Novel Modulator of Oxidative Phosphorylation on Kidney Function in Patients With Progressive Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Neukidney Inc. (Industry)
Responsible Party: Principal Investigator, Ebima Clifford Okundaye, Principal investigator, Neukidney Inc.
Other Study IDs: 0001A
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease (Stage 3-4); Chronic Kidney Disease (Stages 4 and 5); Proteinuria
Keywords: CKD; CHRONIC KIDNEY; KIDNEY DISEASE; KIDNEY DECLINE; PROGRESSION OF CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with progressive chronic kidney disease: GFR decline
  Interventions: Drug: QRX-3; Drug: Eseronate

INTERVENTIONS:
Drug: QRX-3 — Compounded new drug regime
Drug: Eseronate — Neukidney innovative drug
  Other Names: QRX-3

SUMMARY:
Outcome of use of a novel Modulator of Oxidative Phosphorylation on kidney function in patients with Chronic Kidney Disease

DETAILED DESCRIPTION:
QRX-3 ( Eseronate ) is a formulated drug designed to supply and optimize NAD+ mitochondrial availability in order to target the loss of nephrons via renal fibrosis and tubular senescence of the kidney cells by enhancing the mitochondrial activity of these cells via the NAD/NAD+ redox pathway as well as reduce the presence of fibrogenic intracellular inflammatory markers . This novel drug therapy stabilized the intracellular oxidative phosphorylation process a pathway mechanism that is dysregulated or abnormal in the ongoing renal tubular cell injury and damage in chronic kidney disease.

In this study the investigators evaluate the effect of intervention with this novel drug therapy on a chronic kidney disease CKD population with slowly progressively declining renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic kidney disease
* Estimated Glomerular function by MDRD of less than 60mls/min
* Patients with declining renal function ( as measured by eGFR by MDRD )
* Rate of decline of eGFR over the last one year of less than 20%
* Negative Serology markers for CKD etiology
* Provider perceived adherence to study follow up

Exclusion Criteria:

* • Rapid rate of decline in kidney function of > 20 % over last one year

  * Symptomatic renal failure
  * Presence of any suspected Acute renal failure superimposed
  * Presence of cast , hematuria, or abnormal urinalysis outside of simple UTI
  * No known reversible cause of renal decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic kidney disease stages 3-5
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Decrease rate of GFR decline | 6 months
  Comparism of percentage and mean change in GFR with time

SECONDARY OUTCOMES:
Effect on proteinuria with time | 6 months
  Rate of change in random urine protein/creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ebima okundaye, MD, Principal Investigator — Neukidney Inc.
Locations (1):
- Premier Kidney clinic, Pasadena, Texas, United States

IPD SHARING:
Plan to Share IPD: No